CLINICAL TRIAL: NCT04958694
Title: Coping and Emotional Development for Adolescents to Reduce Stress for Adolescents
Brief Title: CEDARS Intervention: A Coping, Emotional Development, & Stress Reduction Intervention
Acronym: CEDARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Nia Heard-Garris, MD, MSc, FAAP, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2021-4642
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior; Stress Reduction; Adverse Childhood Experiences; Positive Attitude
Keywords: Adolescent Behavior; Stress Reduction; Adverse Childhood Experiences (ACEs); CEDARS; Positive Affect Intervention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Masking Description: Wait-list control, no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEDARS- Active Intervention (Experimental): Using an adapted stress-reduction intervention called the CEDARS, the investigators will pilot the intervention in adolescents (N=20) to determine the feasibility and acceptability of CEDARS implementation and to investigate adolescent stress reduction.
  Interventions: Behavioral: CEDARS
- CEDARS- Waitlisted Control (Other): The investigators will use a wait-listed control for the pilot intervention in adolescents (N=20) to determine the feasibility and acceptability of CEDARS implementation and to investigate adolescent stress reduction.
  Interventions: Behavioral: CEDARS

INTERVENTIONS:
Behavioral: CEDARS — This intervention is intended to help adolescents cope with stress and improve positive affect.

SUMMARY:
Using an adapted stress-reduction intervention called the CEDARS, the investigators will pilot the intervention in adolescents (N=40) to determine the feasibility and acceptability of CEDARS implementation and to investigate adolescent stress reduction. As an exploratory aim, the investigators will explore the influence of the CEDARS on CMH-related behaviors and CMH. The investigators expect that those adolescents who undergo the intervention will have the greatest improvement in mental health symptoms than their waitlisted counterparts. Our secondary hypothesis is that those who report more adversity will also report greater improvement in mental health symptoms than their peers.

DETAILED DESCRIPTION:
This intervention has been adapted based on feedback from previous focus groups with adolescents, clinical staff, community stakeholders, and a CEDARS workgroup.

Participants will be divided into two groups - 20 in the intervention group and 20 in the waitlisted group.

Adolescents in the intervention group will participate in 7 weekly, 1-hour sessions. This online intervention will feature positive affect and stress reduction skills delivered via self-paced and self-guided modules. The skills are taught through brief didactic and semi-interactive videos followed by invitations and opportunities for practice within the session and at home. Participants will complete a baseline, mid-point, and post-intervention survey to determine the influence of the intervention.

There will be one follow-up survey with participants after the intervention. The survey will take place 1 month after the program has concluded.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 14-19
* Adolescents able to speak and understand English fluently
* Adolescents with reliable internet access (for virtual access to online modules)

Exclusion Criteria:

* Individuals younger than age 14 and older than age 19
* Individuals who are not able to speak or understand English fluently
* Individuals without reliable internet access

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
CEDARS Intervention | 8 Weeks
  Participants will directly benefit from taking part in the interventions by learning and putting into practice new tools to reduce and manage their stress.
Baseline, Midpoint, and Post-Intervention Surveys | 8 weeks
  Participants will complete a baseline survey, a mid-point survey, and a post-intervention survey (after the completion of the last CEDARS online module).
Post-Intervention Follow-Up | 4 weeks
  There will be one follow-up survey with participants. The final survey will be 1 month post-intervention survey.

CONTACTS AND LOCATIONS:
Overall Officials: Nia Heard-Garris, MD,MSc,FAAP, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided